CLINICAL TRIAL: NCT02947087
Title: Alpha-1 Antitrypsin (AAT) Enhances Islet Autograft Survival
Brief Title: Alpha-1 Antitrypsin (AAT) Enhances Islet Autograft Survival in Patients With Chronic Pancreatitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Hongjun Wang, Professor of Surgery, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Pro00053906; 5R01DK105183 (NIH)
Record Dates: First submitted 2016-10-18; First posted 2016-10-27 (Estimated); Results first posted 2023-05-09 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Chronic Pancreatitis
Keywords: Islet autotransplantation; Alpha1 anti trypsin
MeSH Terms: conditions — Pancreatitis, Chronic; alpha 1-Antitrypsin Deficiency | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prolastin-C (Active Comparator): Subjects will be given Prolastin-C intravenously at 60mg/kg weekly for 4 weeks.
  Interventions: Drug: Prolastin-C
- Placebo (Placebo Comparator): Subjects will be given Saline weekly for 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Prolastin-C — Patients will receive Prolastin-C at 60mg/kg on day 0, 7, 14, and 21 days of transplantation
  Other Names: AAT
  Arms: Prolastin-C
Drug: Placebo — Patients will receive saline on day 0, 7, 14, and 21 days of transplantation
  Other Names: Saline
  Arms: Placebo

SUMMARY:
Primary objective: To describe and compare the safety and efficacy of treatment with AAT in chronic pancreatitis patients who undergo total pancreatectomy and islet autotransplantation (TP-IAT).

DETAILED DESCRIPTION:
The goal of this study is to assess whether infusion of Prolastin-C during peri-transplant period can enhance islet autograft survival and function in chronic pancreatitis patients who have total pancreatectomy and islet autotransplantation. This is a prospective, controlled, double-blind study. The primary endpoint will be area under the curve for the serum C-peptide level during the first 4 hours of an mixed meal tolerance test (MMTT), normalized by the number of islet equivalents (IEQ)/kg at day 365±14 after the transplant.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for total pancreatectomy and islet auto-transplantation
* Age > 18 years
* Diabetes free before surgery

Exclusion Criteria:

* Patients who are under immunosuppression
* Patients who have had Puestow or Frey pancreatic surgery
* Patients who have Immunoglobulin A (IgA) deficiency, known antibodies against IgA, or individuals with a history of severe immediate hypersensitivity reactions, including anaphylaxis to Alpha1-proteinase inhibitor products (allergic to AAT)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-01-11 (Actual); Primary Completion 2021-11-13 (Actual); Study Completion 2022-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hongjun Wang, Ph.D, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified dataset available for sharing with researchers
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Available 01MAR2023 indefinitely
Access Criteria: email to Wangho@musc.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prolastin-C | Placebo
Started | 32 | 16
Completed | 29 | 14
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 3 | 2

BASELINE CHARACTERISTICS:
Population: All randomized participants who received total pancreatectomy with islet autotransplantation
Groups:
- Total: Total of all reporting groups
Arm/Group | Prolastin-C | Placebo | Total
Number analyzed (Participants) | 29 | 14 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 14 | 43
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 10 | 28
  Male | 11 | 4 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 29 | 13 | 42
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 26 | 14 | 40
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 29 | 14 | 43

OUTCOME MEASURES:

1. Primary Outcome: Islet Graft Function
Description: Islet graft function will be measured by 4 hour mixed meal tolerance test (MMTT) at 365 days post transplantation. Specific measurement is the C-peptide area under the curve (AUC)
Time Frame: 365 days
Population: All consented participants who received TPIAT
Measure: Mean (Standard Error); unit: ng/ml*min
Arm/Group | Prolastin-C | Placebo
Number analyzed (Participants) | 29 | 14
ng/ml*min | 233 (42) | 354 (78)

ADVERSE EVENTS:
Time Frame: 1 year
Description: Adverse events affecting >3% of the study population and all Serious Adverse Events were collected for 1 year after total pancreatectomy and included time during hospital stays. All participants had chronic abdominal pain at baseline that was prompting frequent hospitalizations. Two participants in the control arm and 3 persons in the MSC arm that withdrew consent and did not get surgery were not included in the adverse event denominator by prospective data safety analysis plan.
Arm/Group | Prolastin-C | Placebo
All-Cause Mortality (participants affected / at risk) | 2/29 | 0/14
Serious Adverse Events (participants affected / at risk) | 22/29 | 8/14
Other Adverse Events (participants affected / at risk) | 15/29 | 6/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prolastin-C (N=29) | Placebo (N=14)
Abdominal Pain (Gastrointestinal disorders) | 10 (13) | 4 (10)
Nausea and Vomitting (Gastrointestinal disorders) | 3 (5) | 2 (6)
Gastric Ulcer with or without bleeding (Gastrointestinal disorders) | 6 (6) | 1 (1)
Colitis (Gastrointestinal disorders) | 3 (4) | 1 (1) — Includes C. difficile colitis and other post surgical causes
Abdominal Fluid Collection (Gastrointestinal disorders) | 3 (4) | 2 (2)
Hyperglycemia (Endocrine disorders) | 2 (2) | 2 (5) — Includes admissions for diabetic ketoacidosis
Portal Vein Thrombosis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Septic Shock (Infections and infestations) | 1 (1) | 0 (0)
GI Bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prolastin-C (N=29) | Placebo (N=14)
Abdominal Pain (Gastrointestinal disorders) | 3 (11) | 3 (3) — Worsening from baseline
Fatigue (General disorders) | 2 (3) | 0 (0)
Nausea and Vomitting (Gastrointestinal disorders) | 1 (1) | 1 (2)
Hypotension (Cardiac disorders) | 3 (3) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Urticaria (Immune system disorders) | 0 (0) | 1 (1)
Hyperglycemia (Endocrine disorders) | 0 (0) | 1 (2)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Portal Vein Thrombosis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Wound seroma (Surgical and medical procedures) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-14): https://cdn.clinicaltrials.gov/large-docs/87/NCT02947087/Prot_SAP_000.pdf